CLINICAL TRIAL: NCT04737642
Title: Feasibility and Safety of Intraoperative Bile Duct Clearance by Sphincter of Oddi Balloon Dilatation: A Prospective Observational Pilot Study
Brief Title: Feasibility and Safety of Bile Duct Clearance by Transcystic Sphincter of Oddi Balloon Dilatation
Acronym: TCPBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BASEC 2020-01066
Record Dates: First submitted 2020-12-24; First posted 2021-02-04 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cholecystolithiasis; Choledocholithiasis; Surgery
MeSH Terms: conditions — Cholecystolithiasis; Choledocholithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Papillary ballon dilatation (Experimental)
  Interventions: Procedure: Papillary ballon dilatation

INTERVENTIONS:
Procedure: Papillary ballon dilatation — Trans cystic papillary ballon dilatation during cholecystectomy

SUMMARY:
To investigate feasibility and safety of intraoperative bile duct clearance by sphincter of Oddi balloon dilatation via cystic duct at cholecystectomy.

Primary endpoint: rate of successful bile duct stone clearance (feasibility). Secondary endpoints (safety): rate of peri-interventional complications (injury to the common bile duct, bleeding, injury to surrounding organs: stomach, duodenum, liver) and short-term postoperative complications (bile leak, cholangitis, lipasaemia, pancreatitis, pneumonia). Duration of procedure. Length of hospital stay.

DETAILED DESCRIPTION:
Standard approach to address common bile duct stones is endoscopic retrograde cholangiography (ERC) with sphincterotomy. Those interventions are performed either before or after gallbladder removal (cholecystectomy), thus, requiring at least two interventions. Moreover, ERC with sphincterotomy is associated with a considerable rate of short and long-term morbidity. The main complications are pancreatitis (2-7%), post sphincterotomy bleeding (1-2%), impaired function of the sphincter with reflux of duodenal content to the bile ducts and a consecutive risk for cholangitis, stone recurrence and even a potential higher risk for cholangiocarcinoma.

The aim of this study is to evaluate an alternative surgical approach of bile duct clearance at the time of cholecystectomy. Literature of this approach is scarce; however, it has shown a trend to lower postoperative complications if compared to ERC. The technique of sphincter of Oddi balloon dilatation and bile duct clearance from stones via cystic duct at cholecystectomy has been described in a few case series. These small case series have shown a good success rate of bile stone clearance and low complication rates when applying the balloon dilation technique for smaller stones.

The investigators have used this technique in selected cases with good success as well. However, the technique needs to be assessed regarding feasibility and safety in a consecutive group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature (Appendix Informed Consent Form)
* Patients ≥ 18 years of age
* Patients with gallbladder stones and known or expected concomitant bile duct stones
* Bile duct stones ≤ 6mm in size measured by intraoperative cholangiography

Exclusion Criteria:

* Women who are pregnant
* Declined consent
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Patients with moderate or severe acute cholangitis
* Patients with moderate or severe pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
Rate of successful bile duct stone clearance (feasibility) | During operation, up to 2 hours
  Intraoperative cholangiogram showing no persistent stones in the common bile duct after the study procedure
Rate of successful bile duct stone clearance (feasibility) | At the 6 week follow up appointment
  Patient not showing any signs of choledocholithiasis (fever, pale stool, dark urine, right upper quadrant pain, elevated cholestasis parameters) at 6 week follow up

SECONDARY OUTCOMES:
Number of patients with injury to common bile duct | During operation, up to 2 hours
  Injury to common bile duct is defined as contrast agent leakage from common bile duct during cholangiography or an obvious lesion.
Intraoperative blood loss | During operation, up to 2 hours
  Measured in ml
Intraoperative blood substitution | During operation, up to 2 hours
  Number of erythrocyte concentrates (275ml each)
Number of patients with lesion to surrounding organs | During operation, up to 2 hours
  stomach, duodenum, liver, small bowel, colon
Number of patients with postoperative bile leak | From operation up to 6 weeks postoperative
  Bile leakage is defined as bilirubin concentration in the drain fluid at least 3 times the serum bilirubin concentration on or after postoperative day 3 or as the need for radiologic or operative intervention resulting from biliary collections or biliary peritonitis
Number of patients with postoperative significant bleeding | From operation up to 6 weeks postoperative
  Significant bleeding is defined as a drop in haemoglobin level > 3 g/dl post-operatively compared with the post-operative baseline level and/or any post-operative transfusion of packed red blood cells for a falling haemoglobin and/or the need for radiological intervention (such as embolization) and/or re-operation to stop bleeding
Number of patients with postoperative cholangitis | From operation up to 6 weeks postoperative
  Cholangitis is defined according to the Tokyo Guidelines 2018 [17]: The guidelines encompass systemic TCPBD-Pilot-Tr ial Version 4.0 of 14.09.2020 Page 29 of 41 inflammation (fever, chills or increased inflammatory markers), cholestasis (jaundice or abnormal liver function tests) and imaging (biliary dilation or evidence of stricture, stone or stent). Diagnosis can be suspected in cases of systemic inflammation and one of the two other parameters. Diagnosis is confirmed if all three parameters are present.
Number of patients with postoperative lipasaemia | 4 hours after the operation
  Lipasaemia is defined as elevation in serum lipase to ten times or greater than the upper limit of normal. It is measured 4 hours after the intervention
Number of patients with postoperative acute pancreatitis | From operation up to 6 weeks postoperative
  The diagnosis of acute pancreatitis is defined by the presence of two of the following three criteria: acute onset of persistent, severe, epigastric pain often radiating to the back, elevation in serum lipase or amylase to three times or greater than the upper limit of normal, and characteristic findings of acute pancreatitis on imaging (contrast-enhanced computed tomography, magnetic resonance imaging, or transabdominal ultrasonography)

CONTACTS AND LOCATIONS:
Overall Officials: Beat Schnüriger, Prof, Principal Investigator — UVCM, Inselspital Bern
Locations (1):
- Inselspital Bern (Department for Visceral Surgery and Medicine), Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prevost GA, Huber C, Schnell B, Candinas D, Wiest R, Schnuriger B. Feasibility and safety of intraoperative bile duct clearance by antegrade transcystic balloon sphincteroplasty: A prospective observational pilot study. J Trauma Acute Care Surg. 2024 Apr 1;96(4):666-673. doi: 10.1097/TA.0000000000004196. Epub 2023 Nov 13. PMID 37962117